CLINICAL TRIAL: NCT05199428
Title: Use of a Deep Phenotyping Platform to Develop a Novel Retinal Imaging Test for Coronary Artery Disease: A Prospective Cross-Sectional Study
Brief Title: Optina Eye to Heart Connection
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Collaborators: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DOC100469
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective cross-sectional, single-center retinal imaging study expecting to enroll approximately 400 male and female subjects ≥ 18 years of age. Subjects having undergone clinically-indicated coronary angiography or coronary computed tomography angiography (CCTA) within one month of consent at the Montreal Heart Institute (MHI) will be screened for inclusion in the study.

DETAILED DESCRIPTION:
This is a prospective cross-sectional, single-center retinal imaging study expecting to enroll aproximately 400 (280 CAD and 120 control) male and female subjects ≥ 18 years of age. Subjects having undergone clinically-indicated invasive coronary angiography or coronary computed tomography angiography (CCTA) within one month of signed consent will be screened for inclusion in the study.

Subjects will be recruited at the Montreal Heart Institute (MHI). During the screening visit, the investigator will review inclusion/exclusion criteria and the following information will be collected: demographic data including age and sex, relevant medical history including risk factors (hypertension, diabetes, dyslipidemia, smoking and obesity), history of CAD, concomitant cardiovascular medications and laboratory tests (lipid profile, fasting glucose) Subjects who provide written informed consent will undergo cognitive evaluation and an ophthalmic examination to identify any ocular exclusion criteria. All eligible subjects will then undergo hyperspectral retinal imaging using a Metabolic Hyperspectral Retinal Camera (MHRC)

Safety will be assessed through reporting of serious adverse events (SAEs) related to retinal imaging procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written informed consent
* Age 18 years or older at the time of informed consent
* Stable (non-emergent) typical or atypical symptoms suspicious for CAD (e.g., chest pain, chest tightness, chest burning, shoulder pain, palpitations, jaw pain, or non-chest pain symptoms such as dyspnea or worsening effort tolerance.
* Patients having undergone clinically-indicated invasive coronary angiography or coronary computed tomography angiography within one month before consent signature

Exclusion Criteria:

1. At Screening Visit 1:

   1. Asymptomatic subjects
   2. Previous coronary revascularization (e.g., coronary artery bypass graft surgery, stenting)
   3. Subjects being evaluated for other cardiac diseases (e.g., valvular disease, cardiomyopathy)
   4. Pregnant or breastfeeding women
2. At Study Visit 2 or Ocular Exclusion Criteria:

   1. Medium or high opacity of the lens
   2. Bleeding in vitreous
   3. Pupillary dilation inadequate or contraindicated
   4. Deficient visual fixation
   5. Refractive error outside of the range -15 to +15
   6. Inability to obtain satisfactory images with the MHRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 400 (280 CAD and 120 control) subjects was chosen to allow for the estimation of the sensitivity and specificity of classification models with an acceptable precision, the latter defined as the corresponding 95% confidence intervals.
  Subjects having undergone clinically-indicated invasive coronary angiography or coronary computed tomography angiography (CCTA) within one month of signed consent will be screened for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of a pre-specified classification model based on retinal imaging parameters | 1.5 year
  Sensitivity and specificity of a pre-specified classification model based on retinal imaging parameters to discriminate between control subjects and subjects with CAD (defined as stenosis in at least one epicardial vessel of 50% or greater) as assessed by coronary angiography.

SECONDARY OUTCOMES:
Correlation between retinal imaging parameters and the number of vessels with a stenosis of 50% or greater as assessed by coronary angiography. | 1.5 year
Correlation between retinal imaging parameters and the maximal severity of coronary artery stenosis as assessed by coronary angiography. | 1.5 year
Sensitivity and specificity of new classification models based on retinal imaging parameters | 1.5 year
  Sensitivity and specificity of new classification models based on retinal imaging parameters to discriminate between control subjects and subjects with CAD (defined as stenosis in at least one epicardial vessel of 50% or greater) as assessed by coronary angiography.
Correlation between retinal imaging parameters and cognitive scores on the Montreal Cognitive Assessment (MoCA) and executive tasks | 1.5 year
Sensitivity and specificity, among CAD subjects, of a pre-specified classification model, as well as new classification models | 1.5 year
  Sensitivity and specificity, among CAD subjects, of a pre-specified classification model, as well as of new classification models, based on retinal imaging parameters to discriminate between subjects with less severe CAD (less vessels with a stenosis of 50% or greater) and subjects with more severe CAD (more vessels with a stenosis of 50% or greater) as assessed by coronary angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardiff, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal heart institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided